CLINICAL TRIAL: NCT02611609
Title: A Phase 1/2 Study to Assess the Safety and Efficacy of MultiStem® Therapy in Subjects With Acute Respiratory Distress Syndrome
Brief Title: A Phase 1/2 Study to Assess MultiStem® Therapy in Acute Respiratory Distress Syndrome
Acronym: MUST-ARDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: Athersys Limited (Industry); Cell Therapy Catapult (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B04-01
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Low dose MultiStem
  Interventions: Biological: MultiStem
- Cohort 2 (Experimental): High dose MultiStem
  Interventions: Biological: MultiStem
- Cohort 3 (Experimental): Highest safe MultiStem dose (from Cohorts 1 and 2) or Placebo
  Interventions: Biological: MultiStem; Biological: Placebo

INTERVENTIONS:
Biological: MultiStem
  Arms: Cohort 1
Biological: MultiStem
  Arms: Cohort 2; Cohort 3
Biological: Placebo
  Arms: Cohort 3

SUMMARY:
A study to examine the safety (and potential efficacy) of the adult stem cell investigational product, MultiStem, in adults who have Acute Respiratory Distress Syndrome (ARDS). The primary hypothesis is that MultiStem will be safe in ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe ARDS, as defined by the Berlin definition, requiring an endotracheal or tracheal tube
* Able to receive investigational medicinal product within 96 hours of meeting the last of the ARDS diagnosis criterion

Exclusion Criteria:

* Concurrent illness that shortens life expectancy to less than 6 months
* Other serious medical or psychiatric illness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Frequency of sustained hypoxemia or hypotension | 4 hours
Suspected Unexpected Serious Adverse Reactions (SUSARs) | 24 hours

SECONDARY OUTCOMES:
Frequency of adverse events | Up to 365 days
Changes in vital signs | Up to 7 days
Changes in blood safety laboratories | Up to 7 days
Ventilator-free days | 28 days
ICU-free days | 28 days
Total length of hospital stay | 28 days
All-cause mortality | 28 days
Changes in levels of oxygenation | Up to 28 days
Changes in positive end-expiratory airway pressure | Up to 28 days
Changes in respiratory physiologic measures including lung compliance and airway resistance (peak and plateau pressures) | Up to Day 365
All-cause mortality | Up to Day 365

OTHER OUTCOMES:
Changes in exploratory blood inflammatory markers | Up to 7 days
Changes in exploratory blood immune markers | Up to 7 days
Quality of Life (QoL) | Up to 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Bellingan, MD, Principal Investigator — University College London Hospital
Locations (10):
- United States (3):
  - University Hospitals - Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - University College London Hospital, London
  - St. Georges Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Bellingan G, Jacono F, Bannard-Smith J, Brealey D, Meyer N, Thickett D, Young D, Bentley A, McVerry BJ, Wunderink RG, Doerschug KC, Summers C, Rojas M, Ting A, Jenkins ED. Safety and efficacy of multipotent adult progenitor cells in acute respiratory distress syndrome (MUST-ARDS): a multicentre, randomised, double-blind, placebo-controlled phase 1/2 trial. Intensive Care Med. 2022 Jan;48(1):36-44. doi: 10.1007/s00134-021-06570-4. Epub 2021 Nov 23. PMID 34811567